CLINICAL TRIAL: NCT03096600
Title: Evaluation of Fast Track Rehabilitaion in Mini-invasive Lombar Arthrodesis
Status: Withdrawn | Type: Observational
Why Stopped: The principal investigator has left the hospital.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: MISS RAL
Record Dates: First submitted 2017-03-26; First posted 2017-03-30 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Rehabilitation
Keywords: spine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mini invasive spine surgery have become very common in the past years. Posterior arthrodesis associated to liberation have good functional results and doesn't present much complication cases.

So that's why St Joseph Hospital spine surgeon have made the hypothesis that this kind of surgery can be associated to fast track surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient accepting fast track réhabilitation for transforaminal lumbar interbody fusion
* age >18 hears

Exclusion Criteria:

* Age >75
* ASA score >2
* long distance between house and hôpital
* socially isolantes
* pathology needed conventional hospitalisation
* psychiatric pathology

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Indications for transforaminal lumbar interbody fusion
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of passage to conventional hospitalization | week 1

SECONDARY OUTCOMES:
Assessment of percentage of patients accepting fast track rehabilitation | day1
Early complication rate | day 30

CONTACTS AND LOCATIONS:
Overall Officials: Pomme JOUFROY, MD, Study Director — GHPSJ

IPD SHARING:
Plan to Share IPD: No